CLINICAL TRIAL: NCT01498900
Title: A Multi-center, Prospective, Non-interventional Evaluation of Efficacy, Safety and Convenience of Using NovoNorm® in the Treatment of Type 2 Diabetic Patients in Routine Clinical Practice
Brief Title: An Observational Study Evaluating Efficacy, Safety and Convenience of NovoNorm® in Treatment of Type 2 Diabetes in Routine Clinical Practice
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: AGEE-1875
Record Dates: First submitted 2011-12-21; First posted 2011-12-26 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — repaglinide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Repaglinide
  Interventions: Drug: repaglinide

INTERVENTIONS:
Drug: repaglinide — Prescription according to the product labelling at the physicians' discretion

SUMMARY:
This study is conducted in Africa and Asia. The aim of this study is to evaluate the efficacy, safety and convenience of using repaglinide (NovoNorm®) in type 2 diabetes management in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Newly diagnosed or not adequately controlled with current therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with type 2 diabetes, newly diagnosed or not adequately controlled on their current therapy, who are treated repaglinide by their physicians in accordance with the approved labeling
Sampling Method: Probability Sample
Enrollment: 30554 (Actual)
Dates: Start 2004-08; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
HbA1c (glycosylated haemoglobin)

SECONDARY OUTCOMES:
Fasting Plasma Glucose (FPG)
Postprandial glucose values
Incidence of hypoglycaemia
Adverse drug reactions (ADR)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Istanbul, Turkey (Türkiye)

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com